CLINICAL TRIAL: NCT03845738
Title: Retrospective Evaluation of Clinical Performance of the Astra Tech Implant System EV When Used in Everyday Practice
Status: Completed | Type: Observational
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: C-AS-18-001
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Dental Implants
Keywords: OsseoSpeed; EV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OsseoSpeed EV implant — The investigational product (OsseoSpeed EV implant) is already included in a restoration in the subject at enrollment, thus this study does not involve the installation of any investigational products.

SUMMARY:
This study is designed as a retrospective, multi-center study. The study population consist of subjects who received one or more OsseoSpeed EV implants during the period January 1st 2015 to December 31st 2016. Two hundred subjects will be enrolled, approximately 25-30 subjects per site. The study includes retrospective data collection from subjects' medical records and data collection from one prospective study visit with a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years at time of implant installation.
* Subject signed and dated the informed consent form.
* Having installed one or more OsseoSpeed EV implants between January 1st 2015 and December 31st 2016.

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, according to Investigator's judgement.
* Subject is not willing to participate in the study or not able to understand the content of the study.
* Involvement in the planning or conduct of the study.
* Simultaneous participation in another clinical study that may interfere with the present study.
* Severe non-compliance to Clinical Investigation Plan (CIP) as judged by the Investigator and/or Dentsply Sirona Implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who received OsseoSpeed EV implants, during January 1st 2015 to December 31st 2016, as part of a prosthetic restoration replacing one or more teeth, in any position in the mouth.
  The results from this study should be representative for the general population, therefore there will be no subject related restrictions regarding which subjects to include in the study population (except that the subjects needs to be at least 18 years old at time of implant installation).
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Vervaeke, MD, Principal Investigator — Centrum voor tandheelkunde Geluwe, Belgium
Locations (7):
- University of Illinois College of Dentistry, Chicago, Illinois, United States
- Centrum voor tandheelkunde Geluwe, Geluwe, Belgium
- Burlington Prosthodontics, Burlington, Canada
- Oral Hammaslääkärit, Helsinki, Finland
- Germany (2):
  - Implantarium Gernsbach, Gernsbach
  - Universitätsklinik Heidelberg, Klinik und Poliklinik für Mund-, Kiefer- und Gesichtschirurgie, Heidelberg
- Hallands sjukhus Halmstad, Department of Oral & Maxillofacial surgery, Halmstad, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject population recruited in this retrospective study consisted of individuals who received OsseoSpeed EV implants between January 1st 2015 and December 31st 2016, as part of a prosthetic restoration replacing one or more teeth in any position of the mouth.
Units Other Than Participants: Implants
Groups:
- OsseoSpeed EV Implant: The investigational product (OsseoSpeed EV implant) was already included in a restoration in the subject at enrollment, thus this study does not involve the installation of any investigational products.
Period: Overall Study
Arm/Group | OsseoSpeed EV Implant
Started (Enrolled/consented) | 208; 385 Implants
Completed (Initiated (completed Visit 1). Included in the PP analysis.) | 208; 385 Implants
Not Completed | 0; 0 Implants

BASELINE CHARACTERISTICS:
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 98
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 39
  Sweden | 18
  Belgium | 31
  United States | 36
  Finland | 10
  Germany | 74
Smoking status [Count of Participants; unit: Participants]
  Non-smoker | 147
  Ex-smoker | 34
  Occasional smoker | 2
  Habitual smoker | 25
Number of implants per subject [Number; unit: Implants]
  1 implant | 113
  2 implants | 52
  3 implants | 21
  4 implants | 14
  5 implants | 2
  6 implants | 4
  7 implants | 1
  8 implants | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Survived Implants at Time of the Follow-up Visit
Description: Survival defined as implant in situ at time of the follow-up visit. Primary analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 385
Implants
  Implant survival - No | 3
  Implant survival - Yes | 382
  Missing | 0

2. Secondary Outcome: Percent of Successful Implants at Time of the Follow-up Visit
Description: Implant success defined as implant in situ at time of the follow-up visit and no Adverse Device Effects (ADEs) related to the implant or adjacent peri-implant tissues reported from the day when the study product(s) was installed until the end of the study. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 385
Implants
  Implant success - No | 7
  Implant success - Yes | 378
  Missing | 0

3. Secondary Outcome: Percent of Successful Prosthetics at Time of the Follow-up Visit
Description: Prosthetic success defined as implant, abutment and restoration in situ at time of the follow-up visit and no Adverse Device Effects (ADEs) related to the reconstruction or adjacent peri-implant tissues reported from the day when the study position(s) was permanently included in a prosthetic restoration until the end of the study. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Number; unit: Prosthetic outcome
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 385
Prosthetic outcome
  Prosthetic success - No | 30
  Prosthetic success - Yes | 354
  Missing | 1

4. Secondary Outcome: Marginal Bone Levels (MBL)
Description: Bone tissue response was evaluated for each investigational position by measuring Marginal Bone Levels (MBL) on the radiographs.
  Intraoral radiographs were used. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set used for analysis of MBL values at follow-up visit. All subjects with available baseline radiographs were included in the baseline MBL analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Groups:
- OsseoSpeed EV Implant - Available Baseline MBL Values: The investigational product (OsseoSpeed EV implant) was already included in a restoration in the subject at enrollment, thus this study does not involve the installation of any investigational products.
  Due to the retrospective design, baseline radiographs were not available for all subjects.
- OsseoSpeed EV Implant - MBL Values Att Follow-up Visit: The investigational product (OsseoSpeed EV implant) was already included in a restoration in the subject at enrollment, thus this study does not involve the installation of any investigational products.
Arm/Group | OsseoSpeed EV Implant - Available Baseline MBL Values | OsseoSpeed EV Implant - MBL Values Att Follow-up Visit
Number analyzed (Participants) | 142 | 208
Number analyzed (Implants) | 263 | 374
mm
  Mesial: number analyzed (Implants) | 262 | 372
  Mesial | 0.2 (0.78) | 0.3 (0.96)
  Distal: number analyzed (Implants) | 261 | 372
  Distal | 0.3 (0.74) | 0.4 (0.87)
  Average | 0.28 (0.67) | 0.38 (0.89)

5. Secondary Outcome: Soft Tissue Response Measured Through Probing Pocket Depth (PPD) at Time of Follow-up Visit
Description: Soft tissue response evaluated by measuring the PPD of each study position. PPD was evaluated using a periodontal probe. PPD was measured as the distance from the mucosal margin to the bottom of the probable pocket in whole millimeters. PPD mean values, and frequencies per depth, were calculated for each study position. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 382
mm | 2.7 (0.84)

6. Secondary Outcome: Soft Tissue Response Measured Through Bleeding on Probing (BoP) at Time of Follow-up Visit
Description: Presence of BoP was evaluated using a periodontal probe. The proportion of surfaces that showed presence of bleeding were calculated and presented for each study implant position. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Number; unit: Number of implants with bleeding
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 382
Number of implants with bleeding | 90

7. Secondary Outcome: Soft Tissue Response Measured Through Presence of Plaque at Time of Follow-up Visit
Description: Plaque was recorded as presence or absence of plaque by visual inspection. The proportion of surfaces that showed presence of plaque were calculated and presented for each study implant position. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Number; unit: Number of implants with plaque
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Implants) | 382
Number of implants with plaque | 63

8. Secondary Outcome: Patient Reported Outcome on Implant Level at Time of Follow-up Visit
Description: Subject satisfaction was evaluated using a short subject questionnaire of each investigational implant position. Subjects were asked to complete a questionnaire to state their opinion about: 1) chewing function and 2) esthetics and 3) overall level of treatment satisfaction.
  For question 1) the scale ranged from Very bad (1), Bad (2), Neither bad or good (3), Good (4), and Very good (5).
  For questions 2) and 3) the scale ranged from Very dissatisfied (1), Dissatisfied (2), Neither dissatisfied nor satisfied (3), Satisfied (4), and Very satisfied (5).
  Authorized investigational site personnel provided the questionnaire during the investigational visit. The subject was instructed to complete it, one per investigational position, and return it for data entry by site personnel into the electronic-Case Report Form (eCRF). The frequencies of each score were calculated for each question and investigational position. Analysis performed on implant level.
Time Frame: Up to 66 months post-procedure.
Population: PP-analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Completed questionnaires
Arm/Group | OsseoSpeed EV Implant
Number analyzed (Participants) | 208
Number analyzed (Completed questionnaires) | 383
score on a scale
  Chewing function (evaluation 1-5) | 4.7 (0.66)
  Esthetics (evaluation 1-5) | 4.7 (0.79)
  Overall level of treatment satisfaction (evaluation 1-5) | 4.8 (0.56)

ADVERSE EVENTS:
Time Frame: Minimum of 2 years of use up to a maximum of around 4½ years of use
Description: The safety objective of this retrospective investigation was to collect all Adverse Device Effects (ADEs) and Serious Adverse Effects (SADEs), i.e., events related to implants, abutment, restoration, or adjacent peri-implant tissues reported from the day when the implant(s) was installed until the end of the investigation (Visit 1). Due to the retrospective design, non-related Adverse Events (AEs) and Serious Adverse Effects (SAEs) have not been collected.
Arm/Group | OsseoSpeed EV Implant
All-Cause Mortality (participants affected / at risk) | 0/208
Serious Adverse Events (participants affected / at risk) | 0/208
Other Adverse Events (participants affected / at risk) | 15/208
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed EV Implant (N=208)
Abutment related (Product Issues) | 1 (1) — Mechanical/technical events related to abutment.
Prosthesis related (Product Issues) | 8 (8) — Mechanical/technical events related to prosthesis.
Peri-implant tissue related (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03845738/Prot_SAP_000.pdf